CLINICAL TRIAL: NCT01227070
Title: Airflow Obstruction and Biomarkers of Airway Inflammation During and Following Acute Exacerbations of Childhood Asthma
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Jason Debley, MD, MPH, Seattle Chidlren's Hospital
Other Study IDs: SCH IRB 11798; IRUSBUPR0055 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Asthma
Keywords: Asthma, hospitalization, children, exhaled nitric oxide, lung function, breath condensate, cysteinyl leukotrienes
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthmatic
- Healthy Control

SUMMARY:
This study is a longitudinal single-center pilot study designed to describe changes in lung function and levels of noninvasive biomarkers of airway inflammation in children ages 6-18 years over two months following hospitalization for an acute exacerbation of asthma. Forty children ages 6-18 years with asthma who are admitted to Children's Hospital and Regional Medical Center (GCRC) for an asthma exacerbation will be enrolled and complete an initial study visit prior to hospital discharge. Children with asthma will be recruited from the inpatient medical unit. During their initial visit subjects will undergo a clinical assessment and perform spirometry to measure lung function. In addition, exhaled nitric oxide (eNO) concentration will be measured and a sample of exhaled breath condensate (eBC) will be collected during 20 minutes of tidal breathing. Breath condensate will be analyzed to determine the concentration of cysteinyl leukotrienes (CysLT), an important mediator of airway inflammation in asthma. Subjects with asthma will return to the GCRC pediatric satellite at Seattle Children's Hospital for follow-up study visits at 1 week, 2 weeks, and 4 weeks following hospital discharge. During follow-up visits subjects will complete a questionnaire regarding symptoms and medication use since the most recent study visit, will perform spirometry, and have eNO concentration measured and breath condensate collected for CysLT analysis.

The aims of this observational study are to:

1. Assess the association of levels of exhaled nitric oxide and cysteinyl leukotrienes in breath condensate with measures of airflow obstruction (FEV1) and asthma symptoms during, and at one, two, and four weeks following hospital discharge for asthma exacerbation.
2. Compare levels of exhaled nitric oxide and cysteinyl leukotrienes in breath condensate from children ages 6-18 years hospitalized for status asthmaticus to levels from age-matched healthy control subjects without asthma.

ELIGIBILITY:
Inclusion Criteria:

Asthma Group

1. At least a one-year history of physician diagnosed asthma
2. Enrollment within 48 hours of hospitalization, and prior to hospital discharge, for an acute asthma exacerbation.
3. Age 6 - 18 years.
4. Birth at ≥ 36 weeks gestation.
5. Ability to perform acceptable and reproducible spirometry meeting American Thoracic Society guidelines.

Control Group

1. Age 6 - 18 years.
2. No prior history of asthma.
3. Birth at ≥ 36 weeks gestation.
4. Ability to perform acceptable and reproducible spirometry meeting American Thoracic Society guidelines.

Exclusion Criteria:

Asthma Group

1. History of daily oral steroid use during the month before treatment for the current exacerbation.
2. Use of a leukotriene antagonist.
3. Birth at ≥ 36 weeks gestation.

Control Group

1. History of asthma or reactive airway disease.
2. History of a prior illness with wheezing.
3. History of chronic cough (daily over the month prior to enrollment).
4. History of allergic rhinitis.
5. History of atopic dermatitis.
6. History of food allergies.
7. A URI or episode of sinusitis within 3 weeks of study entry.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children ages 6-18 years hospitalized for an asthmat exacerbation, similar aged healthy control children
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
FEV1 | 1 month

SECONDARY OUTCOMES:
FEF25-75 | 1 month
exhaled nitric oxide concentration | 1 month
Breath condensate cysteinyl leukotriene concentration | 1 month
albuterol use | 1 month
school absence | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Debley, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States